CLINICAL TRIAL: NCT04990596
Title: Mechanisms fo Clopidogrel Resistance in Older Adults
Brief Title: Mechanisms fo Clopidogrel Resistance in Older Adults (CEPAGE)
Acronym: CEPAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_9831_CEPAGE
Record Dates: First submitted 2021-05-06; First posted 2021-08-04 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Drug Resistance
Keywords: clopidogrel; primary or secondary prevention of cardiovascular events; older adults; clopidogrel resistance; Drug resistance; Antiplatelet resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Centralized determination of clopidogrel and active metabolite (pharmacology Samples) Centralized determination of plasma markers of platelet activation (hematology Samples) Centralized study of genetic polymorphisms (pharmacology Samples)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Age Group 50 to 59: Inclusion criteria :
  * age 50-100 years old,
  * in consultation or hospitalization in one of the participating centres,
  * treatment with clopidogrel 75 milligrammes per day, for at least 10 days, for primary or secondary prevention of cardiovascular events.
  Non-inclusion criteria :
  * treatment with another antithrombotic drug,
  * myeloproliferative syndrome,
  * platelet count < 100 gigas/liter,
  * acute inflammatory situation: severe sepsis, documented acute infection, chronic systemic inflammatory disease or active cancer,
  * dialysis.
  Interventions: Biological: additional blood sample
- Age Group 60 to 69: Inclusion criteria :
  * age 50-100 years old,
  * in consultation or hospitalization in one of the participating centres,
  * treatment with clopidogrel 75 milligrammes per day, for at least 10 days, for primary or secondary prevention of cardiovascular events.
  Non-inclusion criteria :
  * treatment with another antithrombotic drug,
  * myeloproliferative syndrome,
  * platelet count < 100 gigas/liter,
  * acute inflammatory situation: severe sepsis, documented acute infection, chronic systemic inflammatory disease or active cancer,
  * dialysis.
  Interventions: Biological: additional blood sample
- Age Group 70 to 79: Inclusion criteria :
  * age 50-100 years old,
  * in consultation or hospitalization in one of the participating centres,
  * treatment with clopidogrel 75 milligrammes per day, for at least 10 days, for primary or secondary prevention of cardiovascular events.
  Non-inclusion criteria :
  * treatment with another antithrombotic drug,
  * myeloproliferative syndrome,
  * platelet count < 100 gigas/liter,
  * acute inflammatory situation: severe sepsis, documented acute infection, chronic systemic inflammatory disease or active cancer,
  * dialysis.
  Interventions: Biological: additional blood sample
- Age Group 80 to 89: Inclusion criteria :
  * age 50-100 years old,
  * in consultation or hospitalization in one of the participating centres,
  * treatment with clopidogrel 75 milligrammes per day, for at least 10 days, for primary or secondary prevention of cardiovascular events.
  Non-inclusion criteria :
  * treatment with another antithrombotic drug,
  * myeloproliferative syndrome,
  * platelet count < 100 gigas/liter,
  * acute inflammatory situation: severe sepsis, documented acute infection, chronic systemic inflammatory disease or active cancer,
  * dialysis.
  Interventions: Biological: additional blood sample
- Age Group 90 to 100: Inclusion criteria :
  * age 50-100 years old,
  * in consultation or hospitalization in one of the participating centres,
  * treatment with clopidogrel 75 milligrammes per day, for at least 10 days, for primary or secondary prevention of cardiovascular events.
  Non-inclusion criteria :
  * treatment with another antithrombotic drug,
  * myeloproliferative syndrome,
  * platelet count < 100 gigas/liter,
  * acute inflammatory situation: severe sepsis, documented acute infection, chronic systemic inflammatory disease or active cancer,
  * dialysis.
  Interventions: Biological: additional blood sample

INTERVENTIONS:
Biological: additional blood sample — One sample per patient will be taken 1 to 3 hours after clopidogrel administration. Four additional tubes of 3 mL each will be collected for the study, for a total volume of 12 mL.

SUMMARY:
A clopidogrel resistance rate of 40-50% has been found in the population over 70 years of age, whereas biological resistance, associated with an increased risk of cardiovascular events, is observed in about 20-30% of younger patients. One hypothesis is that the active metabolite is less available in resistant patients. Indeed, 85% of the absorbed clopidogrel undergoes inactivation by esterases. Then the remaining fraction undergoes two steps of metabolisation to the active thiol metabolite by CYP450, essentially the isoform 2C19. In older adults, increased esterase activity and/or decreased CYP450 2C19 activity may lead to a decreased concentration of the active metabolite. Multiple chronic conditions and polypharmacy encountered in older individuals are associated with basal platelet hyperactivity, and may also contribute to a poor response to clopidogrel. No data on the relationship between platelet response and circulating metabolite levels, or on the determinants of response to clopidogrel, are currently available in the geriatric population. Therefore, we propose to analyse the relationship between age and platelet and extra-platelet mechanisms potentially involved in the variability of response to clopidogrel.

DETAILED DESCRIPTION:
This study is a prospective observational multi-centre study. The main objective is assessing the pharmacokinetics (PK) and pharmacodynamics (PD) correlation of clopidogrel action in older adults, i.e. correlation between clopidogrel active metabolite concentration (PK) and platelet response phenotype (PD). The primary outcome is the correlation between the concentration of active metabolite of clopidogrel (PK) over the percentage of maximum aggregation at 10 μM ADP (PD) as a function of age. Inclusion criteria are: age 50-100 years old, hospitalization in one of the 4 participating centres, treatment with clopidogrel 75 milligrammes per day, for at least 10 days. The statistical analysis is a multiple linear regression model with the introduction of an interaction term. The first variable of interest (explanatory) is the concentration of the metabolite. A linear regression model will be used to estimate the proportion of variance explained. The analyses will be conducted with SAS version 9.4 (SAS Institute Inc., Cary, N.C., USA). Results will be published in an international scientific review.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients per 10-year age range, (20 patients per age range from 50 to 100 years included) :

* in consultation or hospitalization in one of the participating centres,
* treatment with clopidogrel 75 mg/d for at least 10 days for primary or secondary prevention of cardiovascular events.
* who have received the information and have not expressed their opposition to participate in the study and who have given their written consent for the performance of genetic examinations and the realization of a biocollection
* affiliated to French social security system

Exclusion criteria :

* treatment with another antithrombotic agent,
* myeloproliferative syndrome,
* platelet count < 100 G/L,
* acute inflammatory situation: severe sepsis, documented acute infection, chronic systemic inflammatory disease or active cancer,
* under dialysis,
* no participation in another clinical study,
* deprived of liberty

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from 50 to 100 years treated with clopidogrel 75 mg/d for at least 10 days for primary or secondary prevention of cardiovascular events
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
PK/PD correlation - clopidogrel active metabolite concentration (pharmacokinetics PK in ) / platelet response phenotype(pharmacodynamics, PD) | Day 0
  Correlation PK (concentration of active metabolite of clopidogrel) / PD (%maximum aggregation at 10 μM ADP) as a function of age

SECONDARY OUTCOMES:
Correlation of prodrug/active metabolite concentrations | Day 0
  Ratio of prodrug/active metabolite concentrations as a function of age
Correlation between the area under the curve of aggregationat 10 μM ADP and the concentration of the active metabolite of clopidogrel | Day 0
  Correlation between the area under the curve of aggregation at 10μM ADP and the concentration of the active metabolite of clopidogrelas a function of age
Correlation between the Platelet Reactivity Index of VASPphosphorylation and the concentration of the active metabolite of clopidogrel | Day 0
  Correlation between the Platelet Reactivity Index of VASP phosphorylation and the concentration of the active metabolite of clopidogrel in relation to age
Determination of factors influencing PK/PD response | Day 0
  clinical data: gender
Determination of factors influencing PK/PD response | Day 0
  clinical data: body mass index in kg/m^2
Determination of factors influencing PK/PD response | Day 0
  clinical data: Cumulative Illness Rating Scale-Geriatric

CONTACTS AND LOCATIONS:
Overall Officials: Dominique SOMME, MD, Pr, Principal Investigator — CHU de Rennes - Service de Gériatrie; Isabelle GOUIN-THIBAULT, MD, PhD, Principal Investigator — CHU de Rennes - Service d'Hématologie Biologique; Eric PAUTAS, MD, Pr, Principal Investigator — Hôpital Charles Foix - Court séjour Gériatrique; Corinne FRERE, MD, Principal Investigator — CHU Pitié-Salpêtrière - Hématologie Biologique; Elena PAILLAUD, MD, Principal Investigator — Hôpital Européen Georges Pompidou, Service de Gériatrie Aiguë,; Pascale GAUSSEM, MD, Pr, Principal Investigator — Hôpital Européen Georges Pompidou - Service d'Hématologie Biologique,; Jean-Guillaume DILLINGER, MD, Principal Investigator — Hôpital Lariboisière - Service de Cardiologie; Virginie SIGURET, MD, Pr, Principal Investigator — Hôpital Lariboisière - Hématologie Biologique
Locations (4):
- France (4):
  - Hôpital Charles Foix, Paris
  - Hôpital Européen Georges Pompidou,, Paris
  - Hôpital Lariboisière, Paris
  - CHU de RENNES, Rennes

IPD SHARING:
Plan to Share IPD: No